CLINICAL TRIAL: NCT04215809
Title: APG-2575CU101, A Phase Ib Study of APG-2575 as a Single Agent or in Combination With Other Therapeutic Agents in Patients With Relapsed and/or Refractory Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Brief Title: Study of APG-2575 as a Single Agent or in Combination With Other Therapeutic Agents for CLL/SLL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575CU101
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: CLL/SLL
MeSH Terms: interventions — Lisaftoclax

STUDY DESIGN:
Intervention Model Description: The dose escalation study of APG-2575 as monotherapy will use the standard 3+3 design. APG-2575 will be taken orally, once daily starting with a ramp-up treatment and will receive the full dose starting on Day 1 of 28-Day-Cycle 1. The starting target dose of APG-2575 is 200 mg (using ramp-up) and will be increased in subsequent cohorts to 400 mg, 600 mg, 800 mg and 1200 mg accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lisaftoclax 400mg (Experimental): Lisaftoclax 400mg ramp up
  Interventions: Drug: Lisaftoclax
- Lisaftoclax 600mg (Experimental): Lisaftoclax 600mg ramp up
  Interventions: Drug: Lisaftoclax
- Lisaftoclax 800mg (Experimental): Lisaftoclax 800mg ramp up
  Interventions: Drug: Lisaftoclax
- Lisaftoclax 1000mg (Experimental): Lisaftoclax 1,000mg ramp up
  Interventions: Drug: Lisaftoclax

INTERVENTIONS:
Drug: Lisaftoclax — Lisaftoclax investigation drug in ramp up dosing

SUMMARY:
Assess the safety and tolerability, identify dose-limiting toxicities (DLT) and determine the maximum tolerated dose (MTD) / recommended phase 2 dose (RP2D) of lisaftoclax.

DETAILED DESCRIPTION:
The study will be conducted in two (2) parts and each part will consist of a ramp-up period, dose escalation and dose expansion portions. The duration of the ramp-up period will depend on the dose schedule being tested and will be conducted for both monotherapy and combination therapy. The ramp-up will consist of treatment with lisaftoclax given once a day starting at 20 mg on Day 1, 50 mg on Day 2, 100 mg on Day 3, 200 mg on Day 4, 400 mg on Day 5¸ 600 mg on Day 6, 800 mg on Day 7, and 1,000 mg on Day 8. Scheduled maximum cohort doses for evaluation will start at 400 mg of lisaftoclax to a maximum of 1000 mg of lisaftoclax. Consequently, patients with a scheduled maximum dose of 200 mg will have a 3-day ramp-up period, those scheduled at 400 mg, a 4-day ramp-up, and those scheduled at 600 mg, a 5-day ramp-up, etc, see Figure 1. Part 1 will study lisaftoclax at different dose levels including 400 mg, 600 mg, 800 mg, and 1,000 mg as monotherapy with dose expansion at RP2D. Part 2 will be combination of lisaftoclax with rituximab or acalabrutinib. Part 2 will be a 3+3 dose escalation of combination lisaftoclax plus rituximab or acalabrutinib. Expansion cohorts at RP2D for the respective combinations will be conducted to further evaluate safety and anticancer activity

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Histologically confirmed chronic lymphocytic leukemia (CLL) or small lymphocytic leukemia (SLL) according to the 2018 international workshop (IW) CLL criteria who must have relapsed or be refractory to at least one prior therapy for CLL/SLL and require treatment by 2018 IWCLL criteria. In addition, lisaftoclax (600 mg) plus acalabrutinib combination cohort may include patients who are: (1) treatment-naïve, or (2) refractory to venetoclax.
3. Eastern Cooperative Oncology Group (ECOG) ≤ 2.
4. Patient must have objectively documented evidence of disease progression prior to study entry such as: escalating lymphocytes count with an increase > 50% over a period of two months or doubling time in less than 6 months; enlarging adenopathy or splenomegaly; increasing cytopenias; clinical B symptoms -night sweats, fatigue, > 1% weight loss in 6 months, fevers > 100.50F for ≥ one month without infection.
5. Adequate bone marrow function independent of growth factor:

   1. Absolute neutrophil count (ANC) ≥1.0× 109/L in patient without bone marrow involvement. This criterion does not apply to patients with bone marrow involvement by CLL/SLL.
   2. Platelets count ≥30 x 109/L (entry platelet count must be independent of transfusion within 7 days of first dose of lisaftoclax).
6. Adequate renal and hepatic function as indicated by:

   1. Serum creatinine ≤1.5×upper limit of normal (ULN); if serum creatinine is >1.5×ULN, creatinine clearance must be ≥ 50 mL/min, calculated using the Cockcroft and Gault formula(140-Age)x mas (kg)/(72x creatinine mg/dL); multiply by 0.85 if female (Cockcroft 1976).
   2. Total bilirubin ≤1.5 x ULN, except patients with known Gilbert's syndrome.
   3. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2.5 x ULN, Alkaline phosphatase<2.5×ULN.
   4. International normalized Ratio (INR), Prothrombin Time (PT) or Activated Partial Thromboplastin time (APTT) ≤1.5×ULN unless the patient is receiving anticoagulant therapy as long as PT or APTT is within therapeutic range of intended use of anticoagulants.
7. Females of childbearing potential (i.e., not postmenopausal for at least 2 years or surgically sterile) must have negative results for pregnancy test performed:

   1. At screening on a serum sample obtained within 14 days prior to the first lisaftoclax administration;
   2. Prior to dosing on a urine sample obtained on the first day of lisaftoclax administration, if it has been >7 days since obtaining the serum pregnancy test results.
8. Females of childbearing potential and non-sterile males must practice at least one of the following methods of birth control with partner(s) throughout the study and for 90 days after discontinuing lisaftoclax:

   1. Total abstinence from sexual intercourse as the preferred lifestyle of the patient; periodic abstinence is not acceptable;
   2. Surgically sterile partner(s); acceptable sterility surgeries are: vasectomy, bilateral tubal ligation, bilateral oophorectomy or hysterectomy
   3. Intrauterine device (IUD);
   4. Double-barrier method (contraceptive sponge, diaphragm or cervical cap with spermicidal fellies or cream AND a condom);
   5. Hormonal contraceptives (oral, parenteral, vaginal ring or transdermal) for at least 3 months prior to lisaftoclax administration. If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to lisaftoclax administration.
9. Male patients must refrain from sperm donation, from initial lisaftoclax administration until 90 days after the last dose of lisaftoclax.
10. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Patient has undergone allogeneic stem cell transplant < 90 days.
2. Patient has active graft-versus-host disease or require immunosuppressive therapy.
3. Patient has undergone CAR-T cell therapy < 30 days.
4. Richter's Syndrome (patients with previously treated Richter's syndrome will be permitted if they are in remission).
5. Prior anti-BCL-2 treatment (except patients who discontinued treatment for reasons other than disease progression and patients in the lisaftoclax plus acalabrutinib cohort).
6. For the acalabrutinib and lisaftoclax combination cohort: (1) Patients who discontinued due to acalabrutinib toxicity (Note: Patients who received a BTK inhibitor therapy may participate whether, or not, they progressed following BTK inhibitor treatment). (2) Patients who require treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, etc.) at study entry. (Patients receiving proton pump inhibitors who switch to H2 receptor antagonists or antacids are eligible for enrollment to this study arm.) (3) Patients who require or are receiving anticoagulation therapy with warfarin or equivalent vitamin K antagonists within 7 days of first dose of the study drug(s).
7. Active pathogen infections including human immunodeficiency virus syndrome (HIV) infection.
8. Active hepatitis B infection, as defined seropositivity for Hep B surface antigen (HBsAg) or known active Hepatitis C infection as determined by Hepatitis C antibody with elevated liver enzymes as defined in the inclusion criteria or any other evidence of active Hepatitis C such as currently on treatment; or active COVID-19 infection. (Patients who have received COVID-19 vaccination will be considered as eligible for the study).
9. Has known central nervous system (CNS) involvement.
10. Prior malignancy that required treatment and has shown recurrence within 2 years of screening (except for non-melanoma skin cancer or adequately treated carcinoma in situ of cervix or breast). Cancer treated within 2 years with curative intent and without recurrence as well as prostate cancer on active surveillance are allowed.
11. Concurrent treatment with any other investigational agent, received biologics (≤28 days), or small molecule targeted therapies (≤5 half-life) or other anti-cancer therapies (including chemotherapy) ≤14 days of first dose of lisaftoclax.
12. Patient is pregnant or breast feeding.
13. Has received the following within 7 days prior to the first dose of lisaftoclax:

    1. Steroid therapy at a dose greater than prednisone 20 mg daily (or equivalent) for anti-neoplastic intent
    2. CYP3A inhibitors such as fluconazole, ketoconazole, and clarithromycin
    3. Potent CYP3A inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort.
14. Radiation within 14 days of study entry.
15. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that have not recovered to ≤ grade 1 or baseline, except alopecia or neuropathy.
16. Failure to recover adequately, as judged by the Investigator, from prior surgical procedures. For example, patients with active wound healing; patients who have had major surgery within 28 days from 1st dose of lisaftoclax.
17. Has a cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea or anginal pain.
18. Unstable angina or myocardial infarction within 3 months of enrollment.
19. QTc interval> 480ms (Bazett or Fredericia formulae) or other remarkable abnormal ECG findings, including second-degree type II atrioventricular block, third-degree atrioventricular block or bradycardia (ventricular rate of less than 50 beats per minute).
20. Unable to swallow capsules or have gastrointestinal conditions that could affect the absorption of lisaftoclax in the opinion of the Investigator.
21. Uncontrolled concurrent illness including, but not limited to: uncontrolled diabetes mellitus, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
22. Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Toxicity Endpoint: dose limiting toxicity (DLT) | 42 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 6 weeks (2 cycles) of study treatment. These will be assessed via CTCAE version 5.0
Maximally tolerated dose (MTD) | 42 days
  MTD will be determined based on DLTs observed during the first 6 weeks (2 cycles) of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (9):
- United States (7):
  - City of Hope, Duarte, California
  - Mayo Clinic, Jacksonville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Novant Health, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Swedish Health, Seattle, Washington
- Australia (2):
  - Princess Alexandria Hospital, Brisbane, Queensland
  - Frankston Private Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Davids MS, Chanan-Khan A, Ailawadhi S, Ivanov V, Usenko G, Nogaieva L, Kryachock I, Muzhychuk I, Perekhrestenko T, Kyselova O, Myasnikov A, Lukavetskyy L, Uspenskaya O, Marlton P, Proydakov A, Borisenkova E, Winter A, Siddiqi T, Lysa T, Bakirov B, Gabrail N, Ganju V, Konstantinova T, Samoilova O, Karpenko O, Osipov I, Mudenda B, Fu T, Chen Z, Liang Z, Mekala DJ, Li M, Glass L, Ahmad M, De A, Shah V, Wang H, Winkler RE, Yang D, Zhai Y. Safety, tolerability, and pharmacokinetics of lisaftoclax (APG-2575)-based therapy in patients with chronic lymphocytic leukemia: Phase 1b/2 study. Med. 2025 Dec 12;6(12):100885. doi: 10.1016/j.medj.2025.100885. Epub 2025 Oct 17. PMID 41109219